CLINICAL TRIAL: NCT06954675
Title: Bacterial Responses to Enteric Alterations After Ketones
Brief Title: Comparison of Microbiome Changes in Healthy Adults Following Ketone Ester Consumption
Acronym: BREAK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 25-43835
Record Dates: First submitted 2025-04-11; First posted 2025-05-01 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Microbiome Analysis
Keywords: Microbiome; Exogenous ketone; Ketone ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 25g Bis-octanoyl-(R)-1,3-butanediol (C8) (Experimental): Participants will receive 25g of the ketone ester bis-octanoyl-(R)-1,3-butanediol (C8) daily.
  Interventions: Dietary Supplement: Exogenous ketone ester

INTERVENTIONS:
Dietary Supplement: Exogenous ketone ester — 25g Bis-octanoyl-(R)-1,3-butanediol (C8)

SUMMARY:
The goal of this observational study is to learn if a ketone ester can improve the content of the gut microbiome. The main questions it aims to answer are:

* Does a ketone ester reduce age-related signatures in the gut microbiome?
* What changes occur in the gut microbiome after consuming a ketone ester?

Participants will:

* Take a ketone ester every day for seven (7) days
* Collect and ship stool samples within seven (7) days before, during, and within seven (7) days after the study period
* Measure their ketone levels with a urine strip every day after having the drink
* Answer questions about their typical diet on a normal day
* Record their symptoms, if any arise

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 18 to 40 years of age, inclusive, at Virtual Visit 1.
* Subject has a self-reported BMI of 18.5 to 39.9 kg/m2 (inclusive) at Virtual Visit 1.
* Subject is willing and able to comply with all study procedures including maintenance of habitual dietary intake, consumption of study product at specified intervals, written questionnaires including study log and beverage tolerability questionnaire (KETQ), habitual exercise and medication and supplement use.
* Subject has an email address and internet access via computer, phone, or other device, and is willing and able to maintain internet access throughout the trial to complete virtual visits via video conference.
* Subject has no health conditions that would prevent them from fulfilling the study requirements as judged by the Study Clinician on the basis of medical history.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study.

Exclusion Criteria:

* Subject is unable to converse in English or Spanish
* Subject is unable to provide informed consent due to cognitive impairment or insufficient English or Spanish language comprehension
* Subject has been hospitalized within 30 days of Virtual Visit 1.
* Subject has a history or presence of uncontrolled and/or clinically active pulmonary, cardiac (e.g. >= New York Heart Association class III), hepatic, renal, endocrine (including type 1 diabetes), hematologic, immunologic, neurologic (e.g., Alzheimer's or Parkinson's diseases), psychiatric (including unstable depression and/or anxiety disorders) or biliary disorders. Stable chronic disease is not an exclusion criterion unless specified.
* Subject has a clinically important gastrointestinal condition that would potentially interfere with the evaluation of the study beverage [e.g., inflammatory bowel disease, irritable bowel syndrome, chronic constipation, severe constipation (in the opinion of the Study Clinician), history of frequent diarrhea, history of surgery for weight loss, gastroparesis, systemic disease that might affect gut motility according to the Study Clinician, reflux requiring daily medication, history of gastrointestinal ulcers or bleeding, celiac disease, and/or clinically important lactose intolerance].
* Subject has a known allergy, intolerance, or sensitivity to any of the ingredients in the study product, including milk protein.
* Subject is undergoing treatment or active surveillance for cancer, or has been diagnosed with cancer in the prior two years, except for non-melanoma skin cancer.
* Subject has recently used antibiotics within 60 days of Virtual Visit 1.
* Subject has extreme dietary habits (e.g., intermittent fasting or time restricted eating, Atkins diet, vegan, very high protein/low carbohydrate or has used weight-loss medications (including over-the-counter medications and/or supplements) or programs within 30 days of Virtual Visit 1.
* Subject has used medications (over-the-counter or prescription) known to influence gastrointestinal function including, but not limited to, opioids, weight loss medications, antidiarrheals, and antispasmodics) within 30 days of Virtual Visit 1.
* Subject has used ketone supplements (ketone salts or esters, and medium chain triglycerides [MCT]) within 30 days of Virtual Visit 1.
* Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded.
* Subject has a condition the Study Clinician believes would interfere with their ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Change in Microbiome Composition | From baseline sampling to final sampling, including intervention period, at 21 days
  Microbiome composition will be defined as the following components: 1) alpha-diversity as calculated by Shannon Index; 2) beta-diversity; and 3) microbial community taxa and gene number.

SECONDARY OUTCOMES:
Acute Tolerability Symptoms related to Product Ingestion | From start to end of intervention at 7 days
  Symptoms will be assessed daily using a standardized Beverage Tolerability Questionnaire (Stubbs et al. J Nutr Health Aging 2024). Symptoms are rated on a scale of mild, moderate, and severe with the following symptoms: 1) gas/flatulence; 2) nausea; 3) vomiting; 4) abdominal cramping; 5) stomach rumbling; 6) burping; 7) reflux/heartburn; 8) diarrhea; 9) headache; and 10) dizziness.

CONTACTS AND LOCATIONS:
Overall Officials: John C Newman, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Wayne and Gladys Valley Center for Vision, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study that will only be used to inform future trial design, no IPD will be shared externally.